CLINICAL TRIAL: NCT01773980
Title: Activating Rural Clinics and Women With Disabilities to Improve Cancer Screening
Brief Title: CROSSROAD II: Activating Rural Clinics and Women With Disabilities to Improve Cancer Screening
Status: Completed | Type: Observational
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00009030
Record Dates: First submitted 2013-01-18; First posted 2013-01-23 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Breast Cancer; Cervical Cancer; Colorectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Patient and Clinic Intervention: The patient intervention consists of a single 90-minute interactive in-person session.
  The Clinic intervention consists of an educational video, an interactive meeting with clinicians and clinic staff, and a facilitated follow-up meeting with clinic staff.
  Interventions: Other: Clinic Intervention; Other: Patient Intervention
- Patient Intervention Only: The patient intervention consists of a single 90-minute interactive in-person session.
  Interventions: Other: Patient Intervention
- Clinic Intervention Only: The Clinic intervention consists of an educational video, an interactive meeting with clinicians and clinic staff, and a facilitated follow-up meeting with clinic staff.
  Interventions: Other: Clinic Intervention
- Neither Clinic nor Patient Intervention: Consists of no intervention

INTERVENTIONS:
Other: Clinic Intervention — The Clinic intervention consists of an educational video, an interactive meeting with clinicians and clinic staff, and a facilitated follow-up meeting with clinic staff.
  Groups: Clinic Intervention Only; Patient and Clinic Intervention
Other: Patient Intervention — The patient intervention consists of a single 90-minute interactive in-person session.
  Groups: Patient Intervention Only; Patient and Clinic Intervention

SUMMARY:
The goal of this project is to develop and pilot test an innovative approach for overcoming barriers to cancer screening among women with physical disabilities (WWD) in rural Oregon. Many studies have shown that people with disabilities receive fewer indicated cancer screening services and are more likely to have poor cancer-related outcomes, such as late stage at diagnosis, compared to those without disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 50-75 at time of screening
* No personal history of breast, cervical or colorectal cancer
* Not being up-to-date with at least one screening test for breast, cervical, and/or colorectal cancer
* Meets the study definition of disability per screening survey OR
* Be a woman who does not meet the definition of disability per screening survey, but has been matched to a participant who does (observation group).

Exclusion Criteria:

* Non female
* Personal history of breast, cervical, or colorectal cancer
* Coming into clinic for an urgent care issue

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinics
Sampling Method: Non-Probability Sample
Enrollment: 1570 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of participants with improved cancer screening | Duration of the study; Up to 1 year
  A 2 x 2 factorial study design will be used to explore individual and combined effects of a clinic-based intervention AND a patient-based intervention on improving breast, cervical and colorectal cancer screening among rural women with physical disabilities (WWD).

CONTACTS AND LOCATIONS:
Overall Officials: David Buckley, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States